CLINICAL TRIAL: NCT01913470
Title: A Pilot Study of Losartan in the Treatment of Pediatric NAFLD
Brief Title: Study of Losartan in the Treatment of NAFLD in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Miriam Vos, MD (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Children's Healthcare of Atlanta (Other)
Responsible Party: Sponsor-Investigator, Miriam Vos, MD, Assistant Professor of Pediatrics, Emory University
Organization: Emory University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00062895; 1R03DK096157-01A1 (NIH); 1R03DK096157-01 (NIH)
Record Dates: First submitted 2013-07-08; First posted 2013-08-01 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: NAFLD
Keywords: NAFLD; Non-alcoholic Fatty Liver Disease; Obesity; Pediatrics; Children; Losartan; Cozaar
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Losartan then Placebo (Experimental): 0.4mg/kg/day (max 25mg) for one week and then increase to 0.8mg/kg/day (max 50mg) for 7 additional weeks then placebo pill for 8 weeks
  Interventions: Drug: Losartan
- Sugar pill (Experimental): placebo pill taken for 8 weeks then 0.4mg/kg/day (max 25mg) for one week and then increase to 0.8mg/kg/day (max 50mg) for 7 additional weeks
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Losartan — Oral tablet to be taken once daily at 0.4mg/kg/day (max 25mg) for one week and then increased to 0.8mg/kg/day (max 50mg) for 7 additional weeks.
  Other Names: Cozaar; Losartan Potassium Tablets; Serial Number: 74193404

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is the most common liver disease among children and is closely associated with obesity and the metabolic syndrome. NAFLD increases risk of mortality and natural history studies of adults show that NAFLD is an independent risk factor for cardiovascular disease. Pediatric NAFLD is particularly concerning from a public health standpoint, as it represents an early and possibly more aggressive form of the disease. Currently there is no effective treatment for pediatric NAFLD.

Losartan is an orally-administered angiotensin II receptor antagonist which is currently on the market to treat high blood pressure. The renin-angiotensin-aldosterone (RAA) system has been shown to be important in many disease states including renal disease, cardiovascular disease, and NAFLD. Angiotensin antagonists are a class of medications that has been proposed as a novel treatment of NAFLD in part because they would treat both the factors increasing cardiovascular (CVD) risks as well as potentially improve steatosis, fibrosis and hepatic inflammation.

This study is a randomized, double-blinded, placebo-controlled pilot study to evaluate whether 8 weeks of Losartan will decrease inflammatory markers among children ages 12-19 with a current diagnosis of NAFLD. Efficacy will be assessed by improvement in alanine aminotransferase (ALT) from baseline. Secondary endpoints will include aspartate aminotransferase (AST), cytokeratin 18 levels, and fasting triglyceride levels among others. Safety will be assessed by the recording of adverse events, clinical laboratory parameters, vital signs and physical examinations.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) > 85th% for age and gender
* History of definite or borderline nonalcoholic steatohepatitis (NASH) diagnosed by liver biopsy using NASH Clinical Research Network (CRN) criteria
* At least 2 months of attempted lifestyle changes after liver biopsy
* Current ALT ≥ 3 times normal (69 U/L for girls, 78 U/L for boys) at enrollment
* Glomerular filtration rate (GRF) > 90
* Weight ≥ 62.5 kg

Exclusion Criteria:

* Other chronic illness requiring daily medication (except medications for mild mental illness, acid reflux, allergies, stable attention deficit hyperactivity disorder (ADHD), or asthma)
* Supplement or anti-oxidant therapy within past 2 weeks
* Renal insufficiency
* Cirrhosis and liver synthetic dysfunction (International Normalized Ratio ≥ 1.5)
* History of hypotension
* Diabetes (or fasting glucose > 125 mg/dL)
* Acute illness within past 2 weeks prior to enrollment (fever > 100.4ºF)
* Pregnancy

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2013-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Vos, MD, MSPH, Principal Investigator — Emory University / Children's Healthcare of Atlanta
Locations (1):
- Emory University / Children's Healthcare of Atlanta, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Vos MB, Jin R, Konomi JV, Cleeton R, Cruz J, Karpen S, Rodriguez DS, Frediani JK, McCracken C, Welsh J. A randomized, controlled, crossover pilot study of losartan for pediatric nonalcoholic fatty liver disease. Pilot Feasibility Stud. 2018 Jun 5;4:109. doi: 10.1186/s40814-018-0306-4. eCollection 2018. PMID 29992039

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children were recruited from the patient population of Children's Healthcare of Atlanta and the Emory Children's Center Clinics.
Pre-assignment Details: Of the 16 individuals who signed the consent form, 4 were found to be ineligible to participate during screening process, resulting in 12 participants who began the study treatment.
Groups:
- Losartan Followed by Placebo: Recipients of treatment with losartan for 8 weeks followed by 8 weeks of treatment with a placebo
- Placebo Followed by Losartan: Recipients of treatment with a placebo for 8 weeks followed by 8 weeks of treatment with losartan.
Period: Overall Study
Arm/Group | Losartan Followed by Placebo | Placebo Followed by Losartan
Started | 5 | 7
Completed | 5 | 4
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all participants who consented to participate in the study and met eligibility criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Losartan Followed by Placebo | Placebo Followed by Losartan | Total
Number analyzed (Participants) | 5 | 7 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 6 | 11
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Alanine Aminotransferase (ALT) From Baseline to End of Treatment (8 Weeks of Treatment)
Description: The principal objective of this blinded, placebo controlled, crossover pilot study is to evaluate whether 8 weeks of losartan in children with nonalcoholic steatohepatitis (NASH) will decrease inflammation as measured by ALT.
Time Frame: Baseline (Weeks 0 and 14), Endpoint (Weeks 8 and 22)
Population: In this blinded, crossover treatment, study participants received losartan or a placebo for 8 weeks, then completed a 6 week washout period before crossing over to the other treatment for 8 weeks. The placebo results for four participants in the losartan followed by placebo arm were not usable due to carry over effects from the active treatment.
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- Losartan: Recipients of treatment with losartan for 8 weeks.
- Placebo: Recipients of treatment with a placebo for 8 weeks.
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 9 | 5
U/L
  ALT at Baseline (weeks 0 and 14) | 136.44 (80.06) | 117.40 (56.42)
  ALT at End of Treatment (weeks 8 and 22) | 112.78 (69.64) | 89.40 (35.26)

2. Secondary Outcome: Change in Cholesterol Levels From Baseline to End of Treatment (8 Weeks of Treatment)
Description: For children, a cholesterol level of less than 170 is considered acceptable, 170-199 is borderline high, and 200 and over is high.
Time Frame: Baseline (Week 0 and 14), End of treatment (Week 8 and 22)
Population: The placebo results for four participants in the losartan followed by placebo arm were not usable due to carry over effects from the active treatment. One additional participant in each treatment group is missing the end of treatment cholesterol level measurement.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 9 | 5
mg/dL
  Cholesterol at baseline (week 0 or 14) | 137.67 (28.81) | 152.80 (18.79)
  Cholesterol at end of treatment (week 8 and/or 22): number analyzed (Participants) | 8 | 4
  Cholesterol at end of treatment (week 8 and/or 22) | 132.38 (23.84) | 144.00 (13.47)

3. Secondary Outcome: Change in Triglyceride Levels From Baseline to End of Treatment (8 Weeks of Treatment)
Description: For children aged 10 to 19, triglyceride levels of less than 90 is considered acceptable, 90 to 129 is borderline high, and greater than or equal to 130 and over is high.
Time Frame: Baseline (Week 0 and 14), End of treatment (Week 8 and 22)
Population: The placebo results for four participants in the losartan followed by placebo arm were not usable due to carry over effects from the active treatment. One participant is missing data for the endpoint measurement of triglyceride levels, following 8 weeks of losartan treatment.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 9 | 5
mg/dL
  Triglyceride at baseline (week 0 or 14) | 97.11 (50.27) | 69.60 (11.87)
  Triglyceride at end of treatment (week 8 or 22): number analyzed (Participants) | 8 | 5
  Triglyceride at end of treatment (week 8 or 22) | 65.75 (25.34) | 80.40 (16.59)

4. Secondary Outcome: Change in Fatty Acid Levels From Baseline to End of Treatment (8 Weeks of Treatment)
Description: In human studies, losartan has been shown to decrease serum free fatty acids, thus any decrease in this measurement indicates a positive response to losartan.
Time Frame: Baseline (Week 0 and 14), End of Treatment (Week 8 and 22)
Population: The placebo results for four participants in the losartan followed by placebo arm were not usable due to carry over effects from the active treatment. One participant is missing the endpoint measurement for free fatty acid levels, following the 8 week losartan treatment phase.
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 9 | 5
mEq/L
  Fatty acid at Baseline (week 0 and 14) | 0.38 (0.17) | 0.41 (0.12)
  Fatty acid at end of treatment (week 8 and 22): number analyzed (Participants) | 8 | 5
  Fatty acid at end of treatment (week 8 and 22) | 0.45 (0.11) | 0.38 (0.12)

5. Secondary Outcome: Changes in Homeostasis Model of Assessment - Insulin Resistance (HOMA-IR) Between Baseline and End of Treatment (8 Weeks of Treatment)
Description: Homeostasis Model of Assessment - Insulin Resistance (HOMA-IR) is an equation which indicates the degree of insulin resistance, where higher scores equate to greater insulin resistance. HOMA-IR is calculated as fasting glucose (mg/dl) × insulin (mU/L)/405. A HOMA-IR value >2.0 in prepubertal children and >2.6 in pubertal children, may be considered a warning sign for pediatricians to further investigate insulin resistance.
Time Frame: Baseline (Week 0 and 14), End of Treatment (Week 8 and 22)
Population: The placebo results for four participants in the losartan followed by placebo arm were not usable due to carry over effects from the active treatment. An additional participant is missing HOMA-IR data from the placebo phase of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 9 | 4
units on a scale
  HOMA-IR at Baseline (week 0 or 14) | 20.12 (11.31) | 6.59 (2.91)
  HOMA-IR at end of treatment (week 8 or 22) | 9.35 (4.81) | 11.67 (4.42)

6. Secondary Outcome: Changes in Plasminogen Activator Inhibitor-1 (PAI-1) Concentrations Between Baseline and End of Treatment
Description: PAI-1 is an acute-phase protein that is associated with both injury and inflammation, and has been found to be elevated in adolescents with significant hepatic steatosis. The reference range for PAI-1 in fasting adults is 3-72 ng/mL
Time Frame: Baseline, Week 8, Week 14, Week 22
Population: The placebo results for four participants in the losartan followed by placebo arm were not usable due to carry over effects from the active treatment. One additional participant is missing PAI-1 data from the placebo phase of the study.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 9 | 4
ng/mL
  PAI-1 at Baseline (week 0 or 14) | 5.25 (1.55) | 6.39 (2.57)
  PAI-1 at end of treatment (week 8 or 22) | 5.04 (2.50) | 6.58 (4.01)

7. Other Pre Specified Outcome: Change in Aspartate Aminotransferase (AST) From Baseline to End of Treatment
Description: The normal range for AST in children is 0 - 60 IU/L. AST can respond rapidly to treatment so decreases between Baseline and subsequent measurements indicate positive effects of treatment.
Time Frame: Baseline, Week 8, Week 14, and Week 22
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 9 | 5
IU/L
  AST at Baseline (week 0 or 14) | 66.89 (28.01) | 51.60 (18.05)
  AST from Baseline to Week 22 | 54.22 (21.52) | 37.80 (10.71)

ADVERSE EVENTS:
Time Frame: Adverse event details were collected throughout the duration of study participation, from the Baseline visit through the Week 28 follow up visit.
Description: For this study, an adverse event is considered any untoward medical occurrence in a subject participating in a clinical study that does not necessarily have a causal relationship with the study drug. It can also mean any unfavorable and unintended sign (including laboratory findings, symptom, or disease) temporarily associated with the use of losartan or placebo, whether or not directly related to losartan or not.
Arm/Group | Losartan | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/5
Other Adverse Events (participants affected / at risk) | 9/9 | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan (N=9) | Placebo (N=5)
Ear ache (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 2 (2) | 0 (0)
Abdominal Pain (General disorders) | 1 (1) | 2 (2)
Chest Pain (General disorders) | 2 (2) | 0 (0)
Dizziness (General disorders) | 3 (4) | 2 (2)
Fatigue (General disorders) | 1 (2) | 0 (0)
Lack of Concentration (General disorders) | 2 (3) | 0 (0)
Nausea (General disorders) | 2 (2) | 2 (2)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 2 (3)
Sinus Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hives (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes